CLINICAL TRIAL: NCT03782181
Title: Randomized Controlled Trial of a Therapeutic Intervention Consisting of the Use of Whole Body Vibration in Patients With Fibromyalgia.
Brief Title: Use of Whole Body Vibration in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IB 2586/15 PI
Record Dates: First submitted 2018-12-16; First posted 2018-12-20 (Actual); Results first posted 2020-01-29 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: In this clinical,two groups of participants receive different interventions. One group receives a training with a whole body vibration plattform and the other is the control group.
Who Masked: Participant, Investigator
Masking Description: In this clinical trial design strategy, the participants and the investigator do not know which participants have been assigned which interventions so there is a double-blind masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration plat (Active Comparator): An arm type in which a group of patients with fibromyalgia receives an intervention based on the use of a whole body vibration platform, considered to be effective by clinical evidence.
  Interventions: Device: Whole body vibration platform
- Control group (No Intervention): No intervention arm

INTERVENTIONS:
Device: Whole body vibration platform — A neuromuscular treatment using a rotational whole body vibration platform.
  Arms: Whole body vibration plat

SUMMARY:
The objective of this study is to evaluate the efficacy of a 3-month program consisted of the use of whole body vibration (WBV) in patients with fibromyalgia in order to determine whether this intervention would be effective to short and medium-term improvement of symptoms in these patients.

DETAILED DESCRIPTION:
This was a single blind randomized controlled trial. Forty patients of FM group were assigned randomly to 2 study groups: 20 patients will be part of the experimental group (EG) that will perform a neuromuscular treatment using the vertical whole body vibration platform and another 20 will constitute the control group (CG). All these subjects will sign the corresponding informed consent for their participation in the study, according to the ethical criteria established in the Helsinki Declaration. The study took place between January and Juny 2019. Two groups of variables were analyzed in the present study three times: before, after and follow-up after three months of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FM were included in the study if they fulfilled the 1990 classification criteria of the American College of Rheumatology for fibromyalgia.
* Pain-free volunteers were included if they did not present pain symptoms or some type of treatment in any part of the body during the previous 12 months.

Exclusion Criteria:

* Participants were excluded from the study if they had not signed the informed consent or if they reported any other musculoskeletal disorder rather than patients with FM, any neurological disorder or had previous spinal fusion surgery or spinal cord stimulation.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José A Mingorance, PhD, Principal Investigator — Balearic Islands University
Locations (1):
- University of Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adsuar JC, Del Pozo-Cruz B, Parraca JA, Olivares PR, Gusi N. Whole body vibration improves the single-leg stance static balance in women with fibromyalgia: a randomized controlled trial. J Sports Med Phys Fitness. 2012 Feb;52(1):85-91. PMID 22327091
- [Result] Sanudo B, de Hoyo M, Carrasco L, Rodriguez-Blanco C, Oliva-Pascual-Vaca A, McVeigh JG. Effect of whole-body vibration exercise on balance in women with fibromyalgia syndrome: a randomized controlled trial. J Altern Complement Med. 2012 Feb;18(2):158-64. doi: 10.1089/acm.2010.0881. Epub 2012 Feb 9. PMID 22321155

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Whole Body Vibration Plat | Control Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is the same from the assignment in participant flow.
Groups:
- Patients Perform Whole Body Vibration Plat: An arm type in which a group of patients with fibromyalgia receives an intervention based on the use of a whole body vibration platform, considered to be effective by clinical evidence.
  Whole body vibration platform: A neuromuscular treatment using a rotational whole body vibration platform.
- Total: Total of all reporting groups
Arm/Group | Patients Perform Whole Body Vibration Plat | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Sex: female or male
  Participants
    Female | 19 | 18 | 37
    Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 20 | 40
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 20 | 20 | 40
weight [Mean (Standard Deviation); unit: kg] | 67 (7.46) | 65 (5.82) | 66 (6.42)

OUTCOME MEASURES:

1. Primary Outcome: Pressure Pain Thresholds
Description: Pressure stimuli were applied on two bilateral body locations: epicondyles and index finger. The pressure pain threshold was defined as the pressure value considered as painful by the participant.
Time Frame: 20 minutes
Population: Patients diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology (n=40).
Measure: Mean (Standard Deviation); unit: Newton/centimeter² (N/cm²)
Groups:
- Whole Body Vibration Plat: An arm type in which a group of patients with fibromyalgia receives an intervention based on the use of a whole body vibration platform, considered to be effective by clinical evidence.
  Whole body vibration platform: A neuromuscular treatment using a rotational whole body vibration platform, on January 18, 2017
Arm/Group | Whole Body Vibration Plat | Control Group
Number analyzed (Participants) | 20 | 20
Newton/centimeter² (N/cm²) | 29.8 (9.7) | 22.1 (6.2)

2. Primary Outcome: Vibration Thresholds
Description: Vibration thresholds at the great toes and at the index fingers were quantified bilaterally using a Vibratron II (Physitemp, Clifton, USA). Using a two-alternative forced-choice procedure, subjects identified which of two rods was vibrating. Vibration values displayed on the control unit are vibration units (the amplitude of vibration, proportional to the square of applied voltage). Vibration threshold for the index finger in the normal population between 18 and 65 years of age is 0.7 vibration units with a standard deviation of 0.4 vibration units. The vibration threshold for the great toe in a similar population is 1.2 vibration units with a standard deviation of 0.5 vibration units. There is an increase in threshold scores and in variance as a function of age. There is an increase in threshold scores and variance depending on age. When the vibratory threshold is lower, it indicates the patient's greater ability to detect vibratory stimuli.
Time Frame: 20 minutes
Population: Patients diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology (n=40).
Measure: Mean (Standard Deviation); unit: Hertz
Arm/Group | Whole Body Vibration Plat | Control Group
Number analyzed (Participants) | 20 | 20
Hertz | 2.8 (0.7) | 3.5 (0.6)

3. Primary Outcome: Berg Scale
Description: This is a functional balance assessment tool, consisting of 14 functional tasks with values ranging from 0 (cannot perform) to 4 (normal performance). The general scores range from 0 (severely impaired balance) to 56 (excellent balance). The Berg scale has been previously used in patients with fibromyalgia to assess balance.
Time Frame: 30 minutes
Population: Patients diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology (n=40).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Whole Body Vibration Plat | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 39.1 (4.8) | 28.4 (3.1)

4. Primary Outcome: Six-minute Walking Test (6MWT)
Description: The 6MWT is a functional test in which the patient walks what he can during 6 minutes, analyzing the total distance walked.
Time Frame: 6 minutes
Population: Patients diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology (n=40).
Measure: Mean (Standard Deviation); unit: Metres
Arm/Group | Whole Body Vibration Plat | Control Group
Number analyzed (Participants) | 20 | 20
Metres | 415 (26.1) | 387 (42.8)

5. Primary Outcome: Dynamometer
Description: A back muscle dynamometer was used to measure isometric back muscle strength.
Time Frame: 5 minutes
Population: Patients diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology (n=40).
Measure: Mean (Standard Deviation); unit: Newtons.
Arm/Group | Whole Body Vibration Plat | Control Group
Number analyzed (Participants) | 20 | 20
Newtons. | 40.8 (5.9) | 32.8 (4.8)

6. Primary Outcome: Analysis of the Romberg's Balance Test With the CvMob Software
Description: The CvMob is an Open Source tool for the movement analysis. The software is capable to analyse the trajectories and to determinate the kinematic variables from a movie, that can be done with a simple camera. The tool includes the Movement Elements Decomposition Method (MED).In the present study, we analyzed the oscillatory body movements during the test performance. These ocillatory movements should be minimal with good balance.The patients were asked to remain in orthostatic position with feet parallel at shoulder height, arms extended along the body and eyes closed for 1 minute. A body marker is placed on the patient's head. A camera placed on the ceiling records the movements. Subsequently, the software analyzes and decomposes the movement that the patient has described in the anteroposterior and mediolateral axis. Higher values represent a worse outcome.
Time Frame: 1 minute
Population: Patients diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology (n=40).
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Whole Body Vibration Plat | Control Group
Number analyzed (Participants) | 20 | 20
Centimeters | 0.004 (0.002) | 0.12 (0.1)

7. Primary Outcome: Gait Task
Description: Subjects were instructed to walk on a 4 meters carpet at their normal walking step, with shocks and with flexed arms positioned on the abdomen. Optical markers were attached at the following three body positions: area between the lateral condyle of the femur and the fibular head, great trochanter and lateral malleolus. Subject's motion was digitally recorded with a video camera at 210 frames per second (CasioExilimEX-FS10). The camera was positioned at a distance of 4 meters from the carpet to visualize changes in position, velocity and anatomical points along the x-axis. It was calculated the stride length by an open- source software for computer vision analysis of human movement.
Time Frame: 5 minutes
Population: Patients diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology (n=40).
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Whole Body Vibration Plat | Control Group
Number analyzed (Participants) | 20 | 20
Meters | 0.9 (0.2) | 1.1 (0.3)

8. Primary Outcome: Fibromyalgia Impact Questionnaire (FIQ)
Description: The Fibromyalgia Impact Questionnaire (FIQ) is an assessment and evaluation instrument developed to measure fibromyalgia (FM) patient status, progress and outcomes. It has been designed to measure the components of health status that are believed to be most affected by fibromyalgia. The FIQ is a self administered instrument that takes approximately 5 minutes to complete. The directions are simple and the scoring is self-explanatory. The FIQ is scored in such a way that a higher score indicates a greater impact of the syndrome on the person. Each of the 10 items has a maximum possible score of 10. Thus the maximum possible score is 100. The average FM patient scores about 50, severely afflicted patients are usually 70 plus.
Time Frame: 5 minutes
Population: Patients diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology (n=40).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Whole Body Vibration Plat | Control Group
Number analyzed (Participants) | 20 | 20
Units on a scale | 69.3 (15.2) | 81.7 (6.6)

9. Primary Outcome: Visual Analogue Pain Scale (VAS)
Description: Each participant was asked to indicate their current level of pain using a 20 cm VAS that ranged from 0 (no pain) to 100 (highest level of pain).
Time Frame: 5 minutes
Population: Patients diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology (n=40).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Whole Body Vibration Plat | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 71.2 (7.9) | 78 (5.2)

10. Primary Outcome: Quality of Life Index (QLI)
Description: The Quality of Life Index (QLI) is a self-report questionnaire that measures perceived health-related quality of life. We used the total score of QLI. Its scale is scored by simply adding the score on each item. The range of scores is between 15 to 105, with a higher score or number being indicative of a higher quality of life. An average total rating for a healthy person is usually around 90, whereas a low quality of life measures around 15.
Time Frame: 10 minutes
Population: Patients diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology (n=40).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Whole Body Vibration Plat | Control Group
Number analyzed (Participants) | 20 | 20
units on a scale | 5.0 (0.9) | 3.8 (0.8)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Whole Body Vibration Plat | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT03782181/Prot_SAP_000.pdf